CLINICAL TRIAL: NCT00674856
Title: A Phase 1 Repeated Dose Open Label Study to Investigate the Pharmacokinetics and Safety of Naproxcinod 750mg Bid Administered to Patients With Impaired Renal Function Compared to Matching Healthy Subjects
Brief Title: A Pharmacokinetics and Safety Study of Naproxcinod in Subjects With Impaired Renal Function
Acronym: HCT3012-X-106
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: NicOx (Industry)
Responsible Party: NicOx, NicOx.
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HCT 3012-X-106
Record Dates: First submitted 2008-05-06; First posted 2008-05-08 (Estimated); Last update posted 2009-01-28 (Estimated); Status verified 2009-01

CONDITIONS: Renal Failure
MeSH Terms: conditions — Renal Insufficiency | interventions — naproxen-n-butyl nitrate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- naproxcinod (Experimental): naproxcinod 750mg(375mg caps x2), administered twice a day.
  Interventions: Drug: naproxcinod

INTERVENTIONS:
Drug: naproxcinod — 750mg

SUMMARY:
To study the pharmacokinetics and safety of naproxcinod in patients with impaired renal function

DETAILED DESCRIPTION:
This is an 8-day, repeated dose, open label study to investigate the pharmacokinetics and safety of naproxcinod in order to guide initial dosing and achieve the optimal dose of naproxcinod in Renal impaired patients.

ELIGIBILITY:
Inclusion Criteria:

* Male or female aged 18 to 75 years with stable mild to moderate renal insufficiency.
* Male or female aged 18 to 75 years with similar distribution of age, weight, gender, smoking habits, and race, and in general good health

Exclusion Criteria:

* Any significant acute or chronic disease (except renal impairment) which may interfere with study evaluations.
* A history of alcohol or drug abuse.
* Diagnosis of gastric or duodenal ulceration and/or history of significant gastro-duodenal bleeding within the last 6 months
* Clinically relevant abnormal ECG
* Current or expected use of anticoagulants or analgesic, anti-inflammatory therapies except low dose aspirin (less than or equal to 325mg per day).
* Participation within 30 days prior to screening in another investigational study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2008-05; Primary Completion 2008-09 (Actual); Study Completion 2008-10 (Actual)

PRIMARY OUTCOMES:
To assess differences in the plasma pharmacokinetics profile of naproxcinod and naproxen (total and unbound) between renal impaired patients and healthy subjects. | 8 days

SECONDARY OUTCOMES:
To assess differences in the plasma and urinary pharmacokinetic profile of naproxcinod metabolites between renal impaired patients and healthy subjects. | 8 days
To assess the general safety of naproxcinod in renal impaired patients and in healthy subjects as shown by the biological tolerance and the adverse events (AE) profile. | 8 days

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Orlando, Florida
  - Minneapolis, Minnesota
  - Saint Paul, Minnesota